CLINICAL TRIAL: NCT01439152
Title: An Open Label Phase I Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Maximum Tolerated Dose of the Anti-mesothelin Antibody Drug Conjugate BAY94-9343 in Subjects With Advanced Solid Tumors
Brief Title: Phase I Study to Determine the Maximum Tolerable Dose of BAY94-9343 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15051; NCT01479335 (obsolete NCT alias)
Record Dates: First submitted 2011-09-01; First posted 2011-09-23 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Oncology
Keywords: Oncology; Solid tumors; Antibody drug conjugate (ADC); Treatment Emergent Adverse Events; Mesothelin
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY94-9343 (Dose-Escalation) (Experimental): BAY94-9343 was administered intravenously in this study. The starting dose for this first-in-man study was 0.15 mg/kg administered as a 1 hour infusion every 21 days. (ENROLLMENT CLOSED).
  Interventions: Drug: BAY94-9343
- BAY94-9343 (Expansion) (Experimental): After Maximum tolerated dose (MTD) had been defined, expansion cohorts were conducted at the MTD dose. Overall up to 32 subjects were planned to be enrolled in the expansion cohort:
  * Ovarian Carcinoma, 20 subjects
  * Mesothelioma, 6-12 subjects (ENROLLMENT CLOSED).
  Interventions: Drug: BAY94-9343 (Expansion)
- BAY94-9343 (1.8 mg/kg) (Experimental): This part of study was randomized and open-label. BAY94-9343 in two parallel dose cohorts of twenty (20) patients with recurrent platinum-resistant or platinum partially-sensitive ovarian cancer and up to four (4) patients with advanced malignant epithelioid peritoneal mesothelioma and eight (8) patients with advanced pleural mesothelioma.
  Interventions: Drug: BAY94-9343 (1.8 mg/kg)
- BAY94-9343 (2.2 mg/kg) (Experimental): This part of study was randomized and open-label. BAY94-9343 in two parallel dose cohorts of twenty (20) patients with recurrent platinum-resistant or platinum partially-sensitive ovarian cancer and up to four (4) patients with advanced malignant epithelioid peritoneal mesothelioma and eight (8) patients with advanced pleural mesothelioma.
  Interventions: Drug: BAY94-9343 (2.2 mg/kg)

INTERVENTIONS:
Drug: BAY94-9343 — BAY94-9343 was administered intravenously in this study. The starting dose for this first-in-man study was 0.15 mg/kg administered as a 1 hour infusion every 21 days.
  Arms: BAY94-9343 (Dose-Escalation)
Drug: BAY94-9343 (Expansion) — BAY94-9343 was administered intravenously in this study. The dose for this expansion cohort was 5.5mg/kg administered as a 1 hour infusion every 21 days.
  Arms: BAY94-9343 (Expansion)
Drug: BAY94-9343 (1.8 mg/kg) — BAY94-9343 was administered intravenously in this study. The dose for this cohort was 1.8 mg/kg administered as a 1 hour infusion every week for 3 weeks.
  Arms: BAY94-9343 (1.8 mg/kg)
Drug: BAY94-9343 (2.2 mg/kg) — BAY94-9343 was administered intravenously in this study. The dose for this cohort was 2.2 mg/kg administered as a 1 hour infusion every week for 3 weeks.
  Arms: BAY94-9343 (2.2 mg/kg)

SUMMARY:
BAY94-9343 was an antibody-drug conjugate (ADC) directed against the cancer antigen mesothelin on tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be ≥ 18 years at the first screening examination / visit
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Life expectancy of at least 12 weeks
* Histologically or cytologically documented invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer (tumors with pseudomyxomatous or mucinous histology are excluded) or advanced predominantly epithelioid peritoneal mesothelioma.

  -- Ovarian cancer must have relapsed >0 months and ≤ 12 months of the prior platinum-based chemotherapy regimen (platinum resistant and partially platinum sensitive).
* All patients must provide the tumor tissue sample [Formalin Fixed Paraffin Embedded (FFPE) slides] from archival tissue or fresh biopsy collected any time before the general screening under the separate informed consent.
* Mesothelin expression in the tumor tissue from archival or fresh biopsy samples defined as the membrane intensity score of 2+ or 3+ (on the 0-3 scale) expressed on at least 30% of tumor cells.

  -- Mesothelin expression must be determined by the validated Investigational Use Only (IUO) assay for ovarian cancer or the prototype immunohistochemistry (IHC) assay for mesothelioma at Ventana at any time before the general screening in patients who had signed a separate informed consent for tumor tissue analysis for mesothelin expression.
* No more than 3 prior lines of systemic cytotoxic therapy for patients with advanced peritoneal or pleural mesothelioma or
* No more than 5 prior lines of systemic cytotoxic therapy for patients with ovarian cancer
* Possible intraperitoneal administration of cytotoxics during surgery will not count as systemic cytotoxic therapy in either case.
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

exclusion Criteria:

* More than 3 prior lines of systemic cytotoxic therapy for patients with advanced peritoneal or pleural mesothelioma
* More than 5 prior lines of systemic cytotoxic therapy for patients with ovarian cancer
* Other systemic anticancer therapies (molecular-targeted, immunotherapy etc.) may be acceptable after the consultation between the Investigator and the Bayer Medical Expert.
* Intraperitoneal administration of cytotoxic anticancer agents during tumor surgery will not count as systemic cytotoxic therapy in this context.
* Prior local radiotherapy is allowed if it is completed at least 4 weeks prior to the first dose of study drug and the subject has evaluable lesions not previously irradiated.
* Anticancer chemotherapy, experimental cancer therapy, or immunotherapy within 2 weeks of start of first dose. Anticancer therapy is defined as any agent or combination of agents with clinically proven anti tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints.
* Radiotherapy to the target lesions within 4 weeks prior to the first BAY94-9343 infusion, if the subject has evaluable tumor lesions not previously irradiated.
* Use of strong inhibitors of P-glycoprotein (transporter) (P-gp) (e.g., ritonavir, cyclosporine, verapamil, and dronedarone) is prohibited from Day -14 and for the duration of the study.
* Impaired cardiac function or clinically significant cardiac disease [i.e., congestive heart failure (CHF) New York Heart Association (NYHA) Class III or IV].
* Left ventriculat ejection fraction (LVEF) <50 % [as measured at screening by Multiple Gated Acquisition scan (MUGA) or echocardiogram].
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management.
* Mild blurry vision, either age-related or due to ocular or systemic disorder (e.g. diabetes, dry eyes, cataracts, uncorrected refraction abnormality) may be allowed at the discretion of the ophthalmologist if deemed as no constituting a predisposition to drug-induced corneal deposits and blurry vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-09-07 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT (dose limiting toxicity) of BAY 94-9343 | At the end of Cycle 1 Day21
Determination of the Pharmacokinetic profile of BAY94-9343 and its metabolites (ADC, Total Antibody, DM4 and DM4-Me) | Cycle 1 and Cycle 3: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, (24), 48, (96), 168, 336 and 504 hours after start of infusion
  Q3W Arm: Cmax, AUC (0-504), AUC (0-tlast), tmax, t1/2 and AUC (Cycle 1 only) Q3W: Cycle 1 and Cycle 3: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, (24), 48, (96), 168, 336 and 504 hours after start of infusion QW Arm:Cmax, AUC(0-168) and tmax) QW: Cycle 1 and Cycle 3: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 24, 48 and 168 hours after start of infusion

SECONDARY OUTCOMES:
Biomarker evaluation: Plasma concentrations of soluble mesothelin and Cytokeratin 18 (CK18) | C1D1: pre-dose, 24, 48, and 168h after start of infusion; C2D1: pre-dose, 4 and 168h after start of infusion; C3D1: pre-dose, 24, 48, and 168h after start of infusion; C4 and every even cycle: pre-dose until Implementation of Am 6
Tumor response: assessment of best response and PFS (progression free survival) according to RECIST (Response Evaluation Criteria in Solid Tumours) 1.1 | 1 year/Screening; Within 5 days before the end of every even cycle until Cycle 8 (Cycle 2, Cycle 4, etc.); Within 5 days before the end of every 4th cycle after Cycle 8 (Cycle 12, 16, etc.); end of treatment
Immunogenicity assessment: assessment of Anti-drug antibody (ADA) formation and neutralizing antibodies (NAs) against anetumab ravtansine | 1 year / Cycle 1, 2 and 3 Day 1: pre-dose; Day 1 of every even cycle starting from Cycle 4 (Cycle 4, 6, 8 etc.): pre-dose until implementation of Am 6
Biomarker evaluation - Levels of mesothelin expression in tumor tissue | Anytime prior to general screening

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- United States (8):
  - New Haven, Connecticut
  - Chicago, Illinois
  - Bethesda, Maryland
  - Detroit, Michigan
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Hassan R, Blumenschein GR Jr, Moore KN, Santin AD, Kindler HL, Nemunaitis JJ, Seward SM, Thomas A, Kim SK, Rajagopalan P, Walter AO, Laurent D, Childs BH, Sarapa N, Elbi C, Bendell JC. First-in-Human, Multicenter, Phase I Dose-Escalation and Expansion Study of Anti-Mesothelin Antibody-Drug Conjugate Anetumab Ravtansine in Advanced or Metastatic Solid Tumors. J Clin Oncol. 2020 Jun 1;38(16):1824-1835. doi: 10.1200/JCO.19.02085. Epub 2020 Mar 26. PMID 32213105